CLINICAL TRIAL: NCT00914095
Title: Study of Methylphenidate to Treat Gait Disorders And Attention Deficit In Parkinson's Disease: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicentric Trial
Brief Title: Study of Methylphenidate to Treat Gait Disorders And Attention Deficit In Parkinson's Disease (PARKGAIT-II)
Acronym: PARKGAIT-II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-005801-20; 2008_25/0832 (Other: sponsor); PHRC 2008/1918 (Other: DHOS); A90135-48 (Other: AFSSAPS)
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2009-06

CONDITIONS: Parkinson's Disease; Gait Disorders, Neurologic; Dementia
Keywords: Parkinson's disease; Freezing of Gait; Methylphenidate; Dopamine transporter inhibitor; Noradrenaline
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic; Dementia | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- methylphenidate (Active Comparator): methylphenidate 10 mg tablets (1 mg /kg /day) 3 time a day
  Interventions: Drug: methylphenidate
- placebo (Placebo Comparator): tablets of placebo 3 time a day
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: methylphenidate — 10 mg tablet of methylphenidate 3 times a day (1 mg/kg/day)
  Other Names: Concerta; Ritaline
  Arms: methylphenidate
Drug: placebo — tablets of placebo 3 times a day
  Arms: placebo

SUMMARY:
Therapeutic management of gait disorders in very advanced Parkinson's disease (PD) patients can sometimes be disappointing, since dopaminergic drug treatments and subthalamic nucleus (STN) stimulation are more effective for limb-related Parkinsonian signs than for gait disorders. Gait disorders could be also partly related to noradrenergic system impairment, pharmacological modulation of both dopamine and noradrenaline pathways could potentially improve the symptomatology. The investigators have demonstrated using an open label study on 17 advanced PD patients that chronic, high doses of methylphenidate (MPD) improved gait, freezing of gait, motor symptoms and attention in the absence of L-Dopa and increased the intensity of response of these symptoms to L-Dopa (Devos et al., 2007). The investigators aimed to confirm their results using a randomized, double-blind, placebo-controlled, parallel-group, multicentric trial. The investigators will assess the clinical value of chronic, high doses (1 mg/kg/day) of MPD vs placebo in 88 non demented PD patients suffering from severe gait disorders with freezing despite their use of optimal dopaminergic doses and eventually STN stimulation parameters. Efficacy will be assessed directly and on video in the absence of L-Dopa and again after acute administration of the drug, both before and after a 3-month course of MPD, using Stand Walk Sit test (primary criteria), the "Freezing Of Gait trajectory", RGSE scale, the UPDRS scores, the dyskinesia rating scale, Achiron scales and using auto-questionnaires of Giladi, ABC scale and PDQ 39. Attention will be assessed using reactions times. Drowsiness will be assessed using Epworth and Parkinson's disease Sleep Scales. Apathy and depression will be monitored with Lille Apathy Rating Scale, MADRS, BPRS, MINI and psychiatric interview. Cardiologic and general tolerance will be also monitored. This study could lead to propose methylphenidate with a good efficacy/ risk balance in advanced PD patients suffering from severe gait disorders with freezing of gait, drowsiness and attention deficit.

DETAILED DESCRIPTION:
Overall study duration: 2 years. Planned inclusion period: 12 months. Study duration for individual patients: 4 months and 2 weeks(2 weeks between screening and randomization, 3 months of double-blind treatment and then a 4-week wash-out period).

Primary objective (V1 and V4):

To assess efficacy of methylphenidate treatment on severe gait disorders including freezing assessed by the Stand Walk Sit Test in patients with advanced Parkinson's disease without dementia or depression and under subthalamic stimulation

Additional Efficacy Endpoints (V1 and V4):

* Gait and motor symptoms: the "Freezing Of Gait trajectory", RGSE scale, the UPDRS scores (partI, II, III, IV), the dyskinesia rating scale
* auto-questionnaires of Giladi, ABC scale and PDQ 39
* Attention: simple and complex reactions times
* Drowsiness: Epworth and Parkinson's disease Sleep Scales
* Apathy Lille Apathy Rating Scale
* Depression and other psychiatric disorders: MADRS, BPRS, MINI and psychiatric interview

Safety and Tolerability Endpoints (V1, V2, V3 and V4):

Tolerability Number of subjects (%) who discontinue the study Number of subjects (%) who discontinue the study due to AEs Safety Measures AE incidence Safety laboratory values Vital signs Blood pressure monitoring ECG Physical and neurological examination

Study Design:

Multicentric study: 12-week double blind, placebo-controlled phase. After being found eligible to participate in the study, subjects will be allocated in a 1:1 ratio into one of the following two treatment groups based on a randomization scheme with blocks stratified:

one methylphenidate

* 1st week: 1/2cp 3 times a day (morning, at noon and at 16h)
* 2nd week: 1cp 3 times a day
* 3rd week: 1cp + 1/2cp 3 times a day
* 4th week: depending on the weight: 2 to 3 cp 3 times a day (1 mg/kg/day)

During the 2 following month: 2 to 3 cp 3 times a day (1 mg/kg/day) one placebo during 3 months same as methylphenidate

Schedule: 10 visits Six short consultations: screening (V0), safety visits every 15 days (V2, V3, V4, V5, V6) and two last consultation for the decrease titration (V8, V9) Two long visits during an hospitalization of two days: randomization (V1, 15 days after V0) and visit of termination (V7, 3 months after randomization)

Patients 76 subjects with Parkinson's disease duration of more than 5 years, without dementia (Mattis Dementia Rating Scale ≥ 130, MMSE ≥ 27 and DSM IV), without major depression (MADRS < 18) who have severe gait disorders including freezing of gait (defined by an answer 2 or 3 at the 3rd question of the autoquestionnaire of Giladi: Do your gait disorders impede your daily living activities and your independence: answer: yes, moderately or severely. But the patient requires no physical assistance to walk) despite an optimal dopaminergic treatment and optimal and if present stable subthalamic stimulation parameters. No additional therapy will be permitted during the study.

Centres :

LILLE :

Neurological department, CHU de Lille, EA 2683, IFR 114 : Pr L. Defebvre, Pr K. Dujardin, Dr D. Devos, Pr Destee, Mme Delliaux. Dr A Kreisler, Dr C Simonin, Dr C. Moreau, Dr A. Delval Department of Pharmacology, Faculté de Médecine, Lille II, EA 1046, IFR 114 : R. Bordet.

CHU AMIENS :Pr. P. KRYSTKOWIAK Place Victor PAUCHET - 80054 AMIENS Cedex 1. CH AIX EN PROVENCE : Dr F. VIALLET Avenue Tamaris - 13616 AIX-en-PROVENCE. APHP - HOPITAL DE LA PITIE SALPETRIERE : Pr M. VIDAILHET 47-83, Boulevard de l'Hôpital - 75 PARIS 13ème CHU BORDEAUX : Pr. F. TISON 1, Avenue Magellan - 33600 PESSAC CHU CLERMONT-FERRANT : Pr. F. DURIF 58, Rue Montalambert - 63000 CLERMONT-FERRRAND CHU CRETEIL : Pr. P. CESARO 51, Avenue du Maréchal de Lattre de Tassigny - 94000 CRETEIL CHU GRENOBLE : Pr P. POLLAK Bd de la Chantourne - BP 217 - 38700 La Tronche. CHU MARSEILLE : Pr. JP AZULAY Hôpital de la Timone - 13385 MARSEILLE cedex 05 CHU NANTES : Pr PH. DAMIER Hôtel-Dieu - Place Alexis Ricordeau - 44093 Nantes cedex 1 CHU POITIERS : Dr JL HOUETO 2, Rue de la Milétrie - 86000 POITIERS. CHU RENNES : Pr. M. VERIN CHU Pontchaillou , Rue H. Le Guilloux - 35033 Cedex 9. CHU ROUEN :DR D. MALTETE

1, Rue Germont - 76000 ROUEN. CHU TOULOUSE : Pr. O. RASCOL Hôpital Purpan - Place du Docteur Baylac - TSA 40031 - 31059 Toulouse cedex 9. CHU STRASBOURG : Pr. C. TRANCHANT Hôpital civil - 1 place de l'hôpital BP 426 - 67091 Strasbourg cedex CHU CAEN : Pr. G. DEFER Avenue Côte de Nacre - 14000 CAEN. CHU NICE : M. BORG Hôpital Pasteur - 30, Avenue de la Voie Romaine - 06000 NICE Promoteur de l'étude : CHRU de Lille

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease of more than 5 years
* Subthalamic nucleus stimulation
* Gait disorders impeding moderately to severely the activities of daily living
* gait disorders including freezing of gait
* able to walk without physical assistance

Exclusion Criteria:

* Dementia (MMSE < 27 et score de Mattis < 130)
* Requiring dopatherapie modification
* Requiring subthalamic stimulation parameters adaptation
* Psychiatric disorders: hallucinations, unstable thymic disorders, psychosis)
* Cardiac disorders: dysrhythmia or unstable arterial hypertension
* Unstable or severe medical illness
* intolerance or contraindication to methylphenidate

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of steps on the Stand Walk Sit Test | 3 months

SECONDARY OUTCOMES:
time on the stand walk sit test | 3 months
number of freezing on the FOG trajectory | 3 months
UPDRS | 3 months
RGSE | 3 months
psychiatric interview | 3 months
Cardiac examination with ECG and blood pressure | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: David Devos, MD, PhD, Principal Investigator — Service de Neurologie, Clinique Neurologique, EA 2683, IFR 114, IMPRT
Locations (1):
- Service de Neurologie, Clinique Neurologique, EA 2683, IFR 114, Lille, France

REFERENCES:
- [Background] Devos D, Krystkowiak P, Clement F, Dujardin K, Cottencin O, Waucquier N, Ajebbar K, Thielemans B, Kroumova M, Duhamel A, Destee A, Bordet R, Defebvre L. Improvement of gait by chronic, high doses of methylphenidate in patients with advanced Parkinson's disease. J Neurol Neurosurg Psychiatry. 2007 May;78(5):470-5. doi: 10.1136/jnnp.2006.100016. Epub 2006 Nov 10. PMID 17098845
- [Derived] Moreau C, Meguig S, Corvol JC, Labreuche J, Vasseur F, Duhamel A, Delval A, Bardyn T, Devedjian JC, Rouaix N, Petyt G, Brefel-Courbon C, Ory-Magne F, Guehl D, Eusebio A, Fraix V, Saulnier PJ, Lagha-Boukbiza O, Durif F, Faighel M, Giordana C, Drapier S, Maltete D, Tranchant C, Houeto JL, Debu B, Azulay JP, Tison F, Destee A, Vidailhet M, Rascol O, Dujardin K, Defebvre L, Bordet R, Sablonniere B, Devos D; Parkgait-II Study Group. Polymorphism of the dopamine transporter type 1 gene modifies the treatment response in Parkinson's disease. Brain. 2015 May;138(Pt 5):1271-83. doi: 10.1093/brain/awv063. Epub 2015 Mar 23. PMID 25805645
- [Derived] Dujardin K, Tard C, Duhamel A, Delval A, Moreau C, Devos D, Defebvre L. The pattern of attentional deficits in Parkinson's disease. Parkinsonism Relat Disord. 2013 Mar;19(3):300-5. doi: 10.1016/j.parkreldis.2012.11.001. Epub 2012 Nov 27. PMID 23196037
- [Derived] Moreau C, Delval A, Defebvre L, Dujardin K, Duhamel A, Petyt G, Vuillaume I, Corvol JC, Brefel-Courbon C, Ory-Magne F, Guehl D, Eusebio A, Fraix V, Saulnier PJ, Lagha-Boukbiza O, Durif F, Faighel M, Giordana C, Drapier S, Maltete D, Tranchant C, Houeto JL, Debu B, Sablonniere B, Azulay JP, Tison F, Rascol O, Vidailhet M, Destee A, Bloem BR, Bordet R, Devos D; Parkgait-II study group. Methylphenidate for gait hypokinesia and freezing in patients with Parkinson's disease undergoing subthalamic stimulation: a multicentre, parallel, randomised, placebo-controlled trial. Lancet Neurol. 2012 Jul;11(7):589-96. doi: 10.1016/S1474-4422(12)70106-0. Epub 2012 Jun 1. PMID 22658702